CLINICAL TRIAL: NCT06372717
Title: A Phase 1 Study to Assess the Safety and Antitumor Activity of APL-4098 Alone and in Combination With Azacitidine and in Combination With Azacitidine Plus Venetoclax in Adults With Acute Myeloid Leukemia (AML), Myelodysplastic Syndrome/AML (MDS/AML) or Myelodysplastic Syndrome With Excess Blasts (MDS-EB)
Brief Title: A Study to Investigate APL-4098 Alone and in Combination in Adults With AML or MDS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Apollo Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP30CP01
Record Dates: First submitted 2024-03-11; First posted 2024-04-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia Refractory; Myelodysplastic Syndrome Acute Myeloid Leukemia; Myelodysplastic Syndrome With Excess Blasts; Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — GATA2 Deficiency; Anemia, Refractory, with Excess of Blasts; Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Escalation Phase: APL-4098 monotherapy (Experimental): Dose escalation with different dosing levels of APL-4098.
  Interventions: Drug: APL-4098
- Dose Escalation Phase: APL-4098 and azacitidine (Experimental): Dose escalation with different dosing levels of APL-4098 in combination with azacitidine.
  Interventions: Drug: Azacitidine and APL-4098
- APL-4098 and azacitidine and venetoclax (Experimental): Dose escalation with different dosing levels of APL-4098 in combination with azacitidine and venetoclax.
  Interventions: Drug: Azacitidine and Venetoclax and APL-4098

INTERVENTIONS:
Drug: APL-4098 — APL-4098 is administered orally in 28-day cycles
  Arms: Dose Escalation Phase: APL-4098 monotherapy
Drug: Azacitidine and APL-4098 — Azacitidine is administered at the standard dose on Day 1 - Day 7 of each 28-day cycle; APL-4098 is administered orally.
  Arms: Dose Escalation Phase: APL-4098 and azacitidine
Drug: Azacitidine and Venetoclax and APL-4098 — Azacitidine is administered at the standard dose on Day 1 - Day 7 of each 28-day cycle; Venetoclax is administered orally; APL-4098 is administered orally.
  Arms: APL-4098 and azacitidine and venetoclax

SUMMARY:
This is an open-label, Phase 1 study to determine the safety, tolerability, and efficacy of APL-4098 alone, and in combination with azacitidine, and in combination with azacitidine plus venetoclax for the treatment of acute myeloid leukemia (AML), myelodysplastic syndrome (MDS)/AML and MDS-excess blasts (EB).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Confirmed diagnosis of relapsed refractory acute myeloid leukemia (R/R AML), myelodysplastic syndrome (MDS)/ AML, or MDS-excess blasts (MDS-EB) with the following characteristics: - R/R AML (primary or secondary, including treatment-related), participant is intolerant to, or considered ineligible for available therapies known to provide clinical benefit.
* WBC count ≤ 25,000/microliter
* ECOG Performance Status of ≤ 2
* Weight ≥ 40kg
* Female participants of childbearing potential must have negative serum pregnancy test at screening; must not plan to become pregnant or have ova harvested or breastfeed while on study; must be willing to use specific contraception or avoid intercourse
* Male participants must be willing to use specific contraception and not plan to impregnant a female partner or donate sperm while on study
* Participant must be willing and able to provide written informed consent and to comply with the requirements of the trial

Exclusion Criteria:

* Certain prior therapies such as: received an allogeneic stem cell transplant within 6 months of screening, received an autologous stem cell transplant within 3 months of screening, received any anti-cancer treatments within 2 weeks of Cycle 1 Day 1, prior radiation therapy within 4 weeks of screening
* Certain medical conditions such as: other malignancies, myocardial infarction within 6 months of screening, symptomatic congestive heart failure, uncontrolled active infection, history of arterial thrombosis within 6 months of screening
* Diagnostic assessments: Left ventricular ejection fraction < 45%, Fridericia's corrected QT interval > 470msec, Aspartate aminotransferase and/or alanine aminotransferase > 3 x upper limit of normal (ULN), total bilirubin > 1.5 x ULN, calculated or measured creatinine clearance < 45 mL/minute (multiply by 0.85 if female)
* Infectious disease: HIV positive, active hepatitis B and/or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events [Safety] | Through study completion, approximately one year
  Evaluation of safety parameters including treatment emergent adverse events as detected by hematology, chemistry, coagulation safety labs, physical exams, vital signs, Electrocardiogram results
Incidence of Dose Limiting Toxicities [Tolerability] | Cycle 1 Day 1 to Cycle 2 Day 1 (a cycle is 28 days)
  Evaluation of tolerability parameters including dose limiting toxicities as detected by hematology, chemistry, coagulation safety labs, physical exams, vital signs, and Electrocardiogram results
Determine Recommended Phase 2 Dose (RP2D)/Recommended dose range (RDR) levels of APL-4098 alone, in combination with azacitidine, and in combination with azacitidine plus venetoclax. | Approximately one year
Assess the Pharmacokinetics of APL-4098 | On Days 1, 2, 8, and 15 of Cycle 1, and on Day 1 of Cycle 2 (each cycle is 28 days)
  Evaluate PK parameters: Maximum plasma concentration (Cmax)
Assess the Pharmacokinetics of APL-4098 | On Days 1, 2, 8, and 15 of Cycle 1, and on Day 1 of Cycle 2 (each cycle is 28 days)
  Evaluate PK parameters: area under the curve (AUC)
Assess the Pharmacokinetics of APL-4098 | On Days 1, 2, 8, and 15 of Cycle 1, and on Day 1 of Cycle 2 (each cycle is 28 days)
  Evaluate PK parameters: Time to peak concentration (Tmax)

SECONDARY OUTCOMES:
Assess response to disease with APL-4098 alone, in combination with azacitidine, and in combination with azacitidine plus venetoclax. | Response is assessed at Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 7 Day 1 (each cycle is 28 days long), then every three cycles thereafter (assessed for up to 2 years)
  R/R AML and MDS/AML participants: response is assessed per European LeukemiaNet (ELN) 2022 criteria MDS-EB participants: response is assessed per revised International Working Group 2023 response criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Aggarwal, MD, Study Chair — Apollo Therapeutics
Locations (7):
- Australia (5):
  - Monash Health, Clayton, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- United Kingdom (2):
  - The Royal Marsden Hospital, London
  - Sarah Cannon Research Institute UK, London

IPD SHARING:
Plan to Share IPD: No